CLINICAL TRIAL: NCT06063681
Title: Phase 1, Dose Escalation, Safety, Tolerability, and Pharmacokinetic Study of SR-8541A (ENPP1 Inhibitor) Administered Orally as Monotherapy or in Combination With Checkpoint Inhibitors in Subjects With Advanced/Metastatic Solid Tumors
Brief Title: A Study of SR-8541A (ENPPI Inhibitor) in Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stingray Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: StingrayTx
Record Dates: First submitted 2023-09-23; First posted 2023-10-02 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-03

CONDITIONS: Advanced / Metastatic Solid Tumor
Keywords: Refractory; Relapsing; Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: The study will follow an accelerated titration dose (ATD) escalation scheme. Single-subject cohorts will open sequentially when previous cohort milestones are met, e.g. completion of the Dose-Limiting Toxicity (DLT) period.
  If the single evaluable subject within an ATD cohort experiences a grade ≥ 2 toxicity during the DLT period, the ATD scheme will stop and a traditional 3+3 design will be implemented.
  The combination part will only commence once the SRC has deemed it safe to proceed and a SR-8541A dose from the dose escalation part is selected as the RP2D. The ICI will be either nivolumab or pembrolizumab and dosing will be per SOC. Both investigational products will start on C1D1. Treatment with ICI may be continued if SR-8541A is discontinued and treatment with SR-8541A may be continued after ICI is discontinued.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SR-8541A Monotherapy (Experimental): SR-8541A will be orally administered.
  Interventions: Drug: SR-8541A; Drug: Immune checkpoint inhibitor (ICI)

INTERVENTIONS:
Drug: SR-8541A — orally administered ENPP1 inhibitor
Drug: Immune checkpoint inhibitor (ICI) — The ICI will be either nivolumab or pembrolizumab.

SUMMARY:
This is an open-label, dose-escalation, multi-center phase 1 study evaluating the safety, tolerability, and pharmacokinetics (PK) of SR-8541A administered orally as a monotherapy or in combination with an immune checkpoint inhibitor (ICI) in subjects with solid tumors.

DETAILED DESCRIPTION:
SR-8541A, an ENPP1 inhibitor, will be administered orally as a monotherapy to assess safety, tolerability, and pharmacokinetics (PK) in subjects with advanced/metastatic solid tumors.

Subjects eligible for treatment include those whose disease is refractory to standard therapeutic options, or for which there are no standard therapeutic options available.

All enrolled patients will orally administer SR-8541A daily. Treatment may continue until the subject's disease worsens or another treatment discontinuation criterion is met.

The combination part will only commence once the SRC has deemed it safe to proceed and a SR-8541A dose from the dose escalation part is selected as the RP2D. The ICI will be either nivolumab or pembrolizumab and dosing will be per SOC. Both investigational products will start on C1D1. Treatment with ICI may be continued if SR-8541A is discontinued and treatment with SR-8541A may be continued after ICI is discontinued.

Approximately 10 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy of at least 3 months
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
3. Histopathologically/cytologically confirmed advanced solid tumor, which is refractory to standard therapeutic options, or for which there are no standard therapeutic options.
4. Measurable disease per RECIST v1.1
5. Willing to provide archival or fresh tumor tissue during screening (required) and post-treatment (optional)
6. Adequate hematologic, renal and hepatic function

Exclusion Criteria:

1. Primary central nervous system (CNS) tumor
2. Prior systemic anti-cancer treatment including other investigational agents, surgery, or radiation within 28 days or 5 half-lives, whichever is less
3. Continuous systemic treatment with either corticosteroids (>10 milligram [mg] daily prednisone equivalents) or other immunosuppressive medications within 28 days
4. Active autoimmune disease that has required systemic treatment in past 2 years
5. History of documented congestive heart failure (New York Heart Association [NYHA] class II - IV); unstable angina; poorly controlled hypertension; clinically significant valvular heart disease; high-risk uncontrolled arrhythmias (including sustained ventricular tachycardia); myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack within the last 6 months, or Canadian Cardiovascular Society angina class > 2
6. Troponin I > ULN
7. Blood pressure (BP) - Systolic < 95 mmHg or > 160 mmHg or diastolic > 100 mmHg
8. Resting heart rate (HR) > 100 beats per minute (BPM)
9. Corrected QT interval by Fridericia (QTcF) ≥ 470 ms
10. Left Ventricular Ejection Fraction (LVEF) < 50%
11. Symptomatic uncontrolled CNS disease requiring treatment with steroids or anti-seizure medications within 2 months
12. Leptomeningeal disease
13. Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for at least 8 weeks
14. Bleeding diathesis due to underlying medical condition or anticoagulation medication which is unable to be promptly reversed by medical treatment
15. Prior additional malignancy that is progressing or has received treatment the previous 3 years
16. Active infection requiring systemic treatment
17. Positive for human immunodeficiency virus (HIV) (HIV antibodies) or active hepatitis B (e.g., HbsAg reactive) or active hepatitis C (e.g., HCV ribonucleic acid [RNA] qualitative) infection with detectable viral load
18. Major surgery within 28 days prior to Day 1 and/or minor surgery (excluding biopsy) within 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events | From first dose of study drug through 30 days following the last dose of study treatment
  Adverse events will be graded according to CTCAE v5.0.
Recommended Phase 2 Dose (RP2D) of SR-8541A | From first dose of study drug through 28 days following the first dose of study treatment
  Based on evaluation of Dose Limiting Toxicities (DLT)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | From first dose of study drug through 28 days following the first dose of study treatment
  Cmax measured in ng/mL
Area under the curve from zero up to time t (AUC0-t) | From first dose of study drug through 28 days following the first dose of study treatment
  AUC0-t measured in ng.h/mL
Area under the concentration time curve from time 0 extrapolated to infinity (AUC0-inf) | From first dose of study drug through 28 days following the first dose of study treatment
  AUC0-inf measured in ng.h/mL
Maximal time for peak concentration (Tmax) | From first dose of study drug through 28 days following the first dose of study treatment
  Tmax measured in h
Terminal phase rate constant (λz) | From first dose of study drug through 28 days following the first dose of study treatment
  λz measured in 1/h
Half-life (t1/2) | From first dose of study drug through 28 days following the first dose of study treatment
  t1/2 measured in h
Overall Response Rate | From first dose of study drug through 2 years following first dose
  Defined as the proportion of subjects in the efficacy population who achieve a radiographic investigator-assessed confirmed complete response (CR)/immune CR (iCR) or partial response (PR)/immune PR (iPR) per RECIST v1.1 or immune Response Evaluation Criteria in Solid Tumors (iRECIST) v1.0
Progression Free Survival | From first dose of study drug through 2 years following first dose
  Defined as the time from start of treatment to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first
Duration of Response | From first dose of study drug through 2 years following first dose
  Defined as the time from the date a response of PR or better was first recorded to the date on which PD was first noted or the date of death due to any cause
Disease Control Rate | From first dose of study drug through 2 years following first dose
  Defined as the proportion of subjects who achieve an investigator-assessed confirmed CR/iCR, PR/iPR, or Stable Disease (SD)/immune SD (iSD) at 16 weeks per RECIST v1.1 or iRECIST v1.0
Overall Survival | From first dose of study drug through 2 years following first dose
  Defined as the time from the start of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Ganju, MD, Principal Investigator — Peninsula & South Eastern Haematology & Oncology Group
Locations (3):
- Australia (3):
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Monash Health, Clayton, Victoria
  - Peninsula & South Eastern Haematology & Oncology Group, Frankston, Victoria

IPD SHARING:
Plan to Share IPD: No